CLINICAL TRIAL: NCT02834247
Title: A Phase 1b Study to Evaluate TAK-659 in Combination With Nivolumab in Patients With Advanced Solid Tumors
Brief Title: A Study of TAK-659 in Combination With Nivolumab in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient efficacy of drug; no safety concern
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C34003; 2016-000853-10 (EudraCT Number); U1111-1181-8312 (Other: WHO)
Record Dates: First submitted 2016-07-12; First posted 2016-07-15 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Triple-Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Head and Neck Carcinoma, Squamous Cell; Advanced Solid Tumors
Keywords: Drug Therapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — TAK-659; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Advanced Solid Tumors (Experimental): TAK-659 60 milligram (mg), tablets, orally, once daily in each 28-day treatment cycle in combination with nivolumab 3 milligram per kilogram (mg/kg), infusion over 60 minutes, intravenously (IV), on Days 1 and 15 in each 28 day treatment cycle until PD or unacceptable toxicity. Dose escalation of TAK-659 to 100 mg may be done using a 3 + 3 dose escalation design to determine a maximum tolerated dose (MTD) and/or RP2D.
  Interventions: Drug: TAK-659; Drug: Nivolumab
- Nivolumab Fixed Dose Cohort (Experimental): After RP2D of TAK-659 has been identified, based on evaluation of combination with weight-based dose of nivolumab (3 mg/kg), RP2D may be evaluated in combination with a fixed dose of 240 mg IV nivolumab after discussion between investigator and sponsor for all types of advanced solid tumors. For single-agent nivolumab, fixed dose is expected to have equal exposure, safety, and efficacy as weight-based (3 mg/kg) dose. If nivolumab fixed dose is evaluated with TAK-659 RP2D, 3 participants will be initially enrolled into cohort. Following evaluation of safety, efficacy, and any available PK data, along with discussions between investigator and sponsor, 3 additional participants may be enrolled into cohort for a total of 3 to 6 participants. If >=1 out of 6 participants experiences dose-limiting toxicity (DLT) in Cycle 1, or significant safety issues are seen in Cycle 2 and beyond, re-evaluation of TAK-659 RP2D when administered with a fixed dose of nivolumab is permitted.
  Interventions: Drug: TAK-659; Drug: Nivolumab
- Part 2: Metastatic Triple-negative Breast Cancer (TNBC) (Experimental): Participants with metastatic TNBC will receive TAK-659 at the RP2D as determined in Part 1, tablets, orally, once daily in each 28-day treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Day 1 and Day 15 of each 28 day treatment cycle until PD or unacceptable toxicity. A subset of participants will receive two weeks of TAK-659 monotherapy during Cycle 1, and will receive nivolumab beginning on Day 15 of Cycle 1. The dose of nivolumab will be either 3 mg/kg or 240 mg IV, dependent on whether the 240 mg fixed-dose cohort is evaluated and deemed safe and tolerable. If so, the dosing regimen may switch to 240 mg, on the basis of change in clinical practice and discussion between the investigator and sponsor. If the nivolumab fixed-dose evaluation cohort is not run, the dose of nivolumab for all participants in the dose expansion phase will be 3 mg/kg.
  Interventions: Drug: TAK-659; Drug: Nivolumab
- Part 2: Metastatic Non-small Cell Lung Cancer (NSCLC) (Experimental): Participants with metastatic NSCLC will receive TAK-659 at the RP2D as determined in Part 1, tablets, orally, once daily in each 28-day treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Day 1 and Day 15 of each 28 day treatment cycle until PD or unacceptable toxicity. A subset of participants will receive two weeks of TAK-659 monotherapy during Cycle 1, and will receive nivolumab beginning on Day 15 of Cycle 1.disease or unacceptable toxicity. The dose of nivolumab will be either 3 mg/kg or 240 mg IV, dependent on whether the 240 mg fixed-dose cohort is evaluated and deemed safe and tolerable. If so, the dosing regimen may switch to 240 mg, on the basis of change in clinical practice and discussion between the investigator and sponsor. If the nivolumab fixed-dose evaluation cohort is not run, the dose of nivolumab for all participants in the dose expansion phase will be 3 mg/kg.
  Interventions: Drug: TAK-659; Drug: Nivolumab
- Part 2: Metastatic HNSCC (Experimental): Participants with Head and Neck Squamous Cell Carcinoma (HNSCC) will receive TAK-659 at the RP2D as determined in Part 1, tablets, orally, once daily in each 28-day treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Day 1 and Day 15 of each 28 day treatment cycle until PD or unacceptable toxicity. A subset of participants will receive two weeks of TAK-659 monotherapy during Cycle 1, and will receive nivolumab beginning on Day 15 of Cycle 1. The dose of nivolumab will be either 3 mg/kg or 240 mg IV, dependent on whether the 240 mg fixed-dose cohort is evaluated and deemed safe and tolerable. If so, the dosing regimen may switch to 240 mg, on the basis of change in clinical practice and discussion between the investigator and sponsor. If the nivolumab fixed-dose evaluation cohort is not run, the dose of nivolumab for all participants in the dose expansion phase will be 3 mg/kg.
  Interventions: Drug: TAK-659; Drug: Nivolumab

INTERVENTIONS:
Drug: TAK-659 — TAK-659 Tablets.
Drug: Nivolumab — Nivolumab intravenous infusion.

SUMMARY:
The purpose of this study is to evaluate the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D), safety and efficacy of TAK-659 in combination with nivolumab in participants with advanced solid tumors.

DETAILED DESCRIPTION:
The drug being tested is TAK-659.This study will look at the determination of the MTD/RP2D and efficacy measured by ORR in participants who take TAK-659 in combination with nivolumab. The study will include a dose escalation phase (Part 1), a potential nivolumab fixed dose cohort, and a dose expansion phase (Part 2).

The study will enroll approximately 120 participants, approximately 9-12 in the dose escalation phase and approximately 36 in each of the 3 dose expansion cohorts. Participants will be assigned to 1 of the 4 treatment groups:

* Part 1: Advanced Solid Tumors
* Potential Nivolumab Fixed Dose Cohort
* Part 2: Metastatic TNBC
* Part 2: Metastatic NSCLC
* Part 2: Metastatic HNSCC

All participants will be asked to take the tablets of TAK-659 at the same time each day throughout the study. Participants will also receive intravenous infusion of nivolumab (within 30 minutes after the TAK-650 dose) once every 2 weeks. This multi-center trial will be conducted globally. The overall time to receive treatment in this study is approximately 12 months. Participants will be assessed for disease response and PD during the PFS follow-up of 6 months (for participants who discontinue due to reasons other than PD) and OS follow-up of 12 months from the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female participant aged 18 years or older.
2. Has eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
3. Female participants who:

   * Are postmenopausal for at least 1 year before the Screening visit, or
   * Are surgically sterile, or
   * If childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participants. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male participants, even if surgically sterilized (that is, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 180 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participants. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
4. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participants at any time without prejudice to future medical care.
5. Suitable venous access for the study-required blood sampling, including PK and pharmacodynamic (PD) sampling.
6. Clinical laboratory values and other measures as specified below within 28 days before the first dose of study drug:

   * Total bilirubin must be <=1.5*the upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be <=2.5*ULN.
   * Creatinine clearance must be greater than or equal to (>=) 60 milliliter per (mL/) minute as estimated by the Cockcroft Gault equation or based on urine collection (12 or 24 hours).
   * Hemoglobin must be >=8 gram per deciliter (g/dL), absolute neutrophil count (ANC) must be >=1500 per microliter (/mcL), and platelet count must be >=75,000/mcL.
   * Lipase must be <=1.5*ULN and amylase <=1.5*ULN with no clinical symptoms suggestive of pancreatitis and cholecystitis.
   * Blood pressure <=Grade 1 (hypertensive participants are permitted if their blood pressure is controlled to <=Grade 1 by hypotensive medications and glycosylated HbA1C <=6.5%).
7. Recovered (that is, <=Grade 1 toxicity) from the reversible effects of prior anticancer therapy.
8. To be enrolled in the dose escalation phase of the study, participants must have a radiographically or clinically evaluable tumor, but measurable disease as defined by RECIST version 1.1 is not required for participation in this study.
9. To be enrolled in the TNBC expansion cohort, participants must have:

   * Histologically confirmed, metastatic TNBC with measurable disease per RECIST version 1.1.
   * Triple-negative disease (estrogen receptor, progesterone receptor, and human epidermal growth factor receptor 2 (HER2) negativity confirmed on a histological biopsy of a metastatic tumor lesion (receptor conversion not allowed).
   * Safely accessible tumor lesions (based on investigator's assessment) for serial pre treatment and post treatment biopsies are required for participants receiving TAK-659 monotherapy run-in treatment for 2 weeks followed by TAK-659 plus nivolumab combination treatment [ approximately 10/30 response-evaluable participants]; adequate, newly obtained, core or excisional biopsy of a metastatic tumor lesion not previously irradiated is required. Mandatory biopsies will be taken before TAK-659 monotherapy, after the 2 weeks of TAK-659 monotherapy, and after 6 weeks of TAK-659 plus nivolumab combination therapy. An optional biopsy may be taken at PD with additional consent from the participants.
   * One, 2, or 3 prior lines of chemotherapy for metastatic disease and with progression of disease on last treatment regimen.
   * For the purposes of this study, neoadjuvant and/or adjuvant chemotherapy regimens do not count as a prior line of therapy.
   * Prior treatment must include an anthracycline and/or a taxane in the neoadjuvant, adjuvant, or metastatic setting with the exception for participants who are clinically contraindicated for these chemotherapies.
10. To be enrolled in the NSCLC expansion cohort, participants must have:

    * Locally advanced or metastatic (stage IIIB, stage IV, or recurrent) NSCLC with measurable lesions per RECIST version 1.1.
    * PD during or following at least 1 prior treatment. Participants should have received a prior platinum-based 2-drug regimen for locally advanced, unresectable/ inoperable or metastatic NSCLC or disease recurrence within 6 months of treatment with a platinum-based adjuvant/neoadjuvant regimen or combined modality (example, chemoradiation) regimen with curative intent.
    * Participants with epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genomic alternations should have PD on prior United States (US) Food and Drug Administration (FDA) approved therapy for these aberrations.
    * Safely accessible tumor lesions (based on investigator's assessment) for serial pretreatment and posttreatment biopsies are required for participants receiving TAK-659 monotherapy run-in treatment for 2 weeks followed by TAK-659 plus nivolumab combination treatment (approximately10/30 response-evaluable participants); adequate, newly obtained, core or excisional biopsy of a metastatic tumor lesion not previously irradiated is required. Mandatory biopsies will be taken before TAK-659 monotherapy, after the 2 weeks of TAK-659 monotherapy, and after 6 weeks of TAK-659 plus nivolumab combination therapy. An optional biopsy may be taken at progression with additional consent from the participants.
11. To be enrolled in the HNSCC expansion cohort, participants must have:

    * Histologically confirmed recurrent or metastatic HNSCC (oral cavity, pharynx, or larynx) that is stage III/IV and not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
    * Histologically confirmed recurrent or metastatic squamous cell carcinoma of unknown primary or nonsquamous histologies (example, mucosal melanoma) are not allowed.
    * Histologically confirmed recurrent or metastatic carcinoma of the nasopharynx is allowed, but these participants will not be included as response-evaluable participants for efficacy analysis of HNSCC.
    * Measurable disease per RECIST version 1.1.
    * Tumor progression or recurrence within 6 months of the last dose of platinum-based therapy in the adjuvant (that is, with radiation after surgery), primary (that is, with radiation), recurrent, or metastatic setting.
    * Safely accessible tumor lesions (based on investigator's assessment) for serial pretreatment and posttreatment biopsies are required for participants receiving TAK-659 monotherapy run-in treatment for 2 weeks followed by TAK-659 plus nivolumab combination treatment (approximately 10/30 response-evaluable participants); adequate, newly obtained, core or excisional biopsy of a metastatic tumor lesion not previously irradiated is required. Mandatory biopsies will be taken before TAK-659 monotherapy, after the 2 weeks of TAK-659 monotherapy, and TAK-659 after 6 weeks of TAK-659 plus nivolumab combination therapy. An optional biopsy may be taken at progression with additional consent from the participants.

Exclusion Criteria:

1. Has active brain metastases or leptomeningeal metastases.
2. Has active, or suspected autoimmune disease or a history of known autoimmune disease, with the exception of:

   o Participants with vitiligo, type I diabetes mellitus, resolved childhood asthma/atopy, residual hypothyroidism due to autoimmune condition requiring only hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
3. Any condition requiring systemic treatment with corticosteroids (less than [>]10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 before first dose of study drug.

   o Corticosteroids for topical use or in nasal spray are allowed, as are inhaled steroids and adrenal replacement steroid doses >10 mg daily in the absence of active autoimmune disease.
4. Has history of pneumonitis requiring treatment with steroids; history of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on the Screening chest computed tomography scan (CT scan); history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
5. Has history of interstitial lung disease.
6. Prior therapy with experimental antitumor vaccines; any T-cell co-stimulation agents or inhibitors of checkpoint pathways, such as anti- programmed cell death protein 1 (PD-1), anti- programmed cell death 1 ligand 1 (PD-L1), anti- programmed cell death 1 ligand 2 (PD-L2), anti-CD137, or anti-CTLA-4 antibody; or other agents specifically targeting T cells are prohibited. However, for dose escalation, prior treatment with the marketed inhibitors of the immune checkpoint pathway, such as nivolumab and pembrolizumab, is allowed. In addition, in each of the expansion cohorts, 6 response-evaluable participants with prior exposure to anti-PD-1 or anti-PD-L1 agents will be allowed to enroll.
7. Has any serious medical or psychiatric illness, including drug or alcohol abuse, that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
8. Has life-threatening illness unrelated to cancer.
9. Is female participant who are lactating and breast-feeding or a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before the first dose of study drug.
10. Systemic anticancer treatment including investigational agents or radiotherapy <2 weeks before the first dose of study treatment (<4 weeks for antibody-based therapy including unconjugated antibody, antibody-drug conjugate, and bi-specific T-cell engager agents; <=8 weeks for cell-based therapy or antitumor vaccine) or have not recovered from acute toxic effects from prior chemotherapy and radiotherapy.
11. Prior treatment with investigational agents =<21 days or =<5*their half-lives (whichever is shorter) before the first dose of study treatment. A minimum of 10 days should elapse from prior therapy to initiating protocol therapy.
12. Major surgery within 14 days before the first dose of study drug and not recovered fully from any complications from surgery.
13. Systemic infection requiring intravenous antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
14. Known human immunodeficiency virus (HIV) positive (testing not required).
15. Known hepatitis B surface antigen-positive or known or suspected active hepatitis C infection (testing not required).
16. Participants with another malignancy within 2 years of study start. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection and are considered disease-free at the time of study entry.
17. Any clinically significant comorbidities, such as uncontrolled pulmonary disease, known impaired cardiac function or clinically significant cardiac disease (specified below), active central nervous system disease, active infection, or any other condition that could compromise the participant's participation in the study.

    Participants with any of the following cardiovascular conditions are excluded:
    * Acute myocardial infarction within 6 months before starting study drug.
    * Current or history of New York Heart Association Class III or IV heart failure
    * Evidence of current uncontrolled cardiovascular conditions including cardiac arrhythmias, angina, pulmonary hypertension, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
    * Fridericia corrected QT interval (QTcF) >450 milliseconds (msec) (men) or >475 msec (women) on a 12-lead electrocardiogram (ECG) during the Screening period.
    * Abnormalities on 12-lead ECG including, but not limited to, changes in rhythm and intervals that in the opinion of the investigator are considered to be clinically significant.
18. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-659 including difficulty swallowing tablets; diarrhea >Grade 1 despite supportive therapy.
19. Use or consumption of any of the following substances:

    * Medications or supplements that are known to be inhibitors of P-glycoprotein (P-gp) and/or strong reversible inhibitors of cytochrome P450 (CYP) 3A within 5 times the inhibitor half-life (if a reasonable half-life estimate is known) or within 7 days (if a reasonable half-life estimate is unknown) before the first dose of study drug. In general, the use of these agents is not permitted during the study.
    * Non-oncology vaccine therapies for prevention of infectious diseases (example, human papillomavirus [HPV] vaccine) within 4 weeks of study drug administration. The inactivated seasonal influenza vaccine can be given to participants before treatment and while on therapy without restriction. Influenza vaccines containing live virus or other clinically indicated vaccinations for infectious diseases (example, pneumovax, varicella) may be permitted but must be discussed with the sponsor's medical monitor and may require a washout period before and after administration of vaccine.
    * Medications or supplements that are known to be strong CYP3A mechanism-based inhibitors or strong CYP3A inducers and/or P-gp inducers within 7 days, or within 5 times the inhibitor or inducer half-life (whichever is longer), before the first dose of study drug. The use of these agents is not permitted during the study.
    * Grapefruit-containing food or beverages within 5 days before the first dose of study drug. Note that grapefruit-containing food and beverages are prohibited during the study.
20. For dose expansion participants who will have tumor biopsies collected:

    * ECOG performance status >1.
    * Activated partial thromboplastin time (aPTT) or plasma thromboplastin (PT) outside the institution's standard of care.
    * Platelet count <75,000/mcL.
    * Known bleeding diathesis or history of abnormal bleeding, or any other known coagulation abnormalities that would contraindicate the tumor biopsy procedure.
    * Ongoing therapy with any anticoagulant or antiplatelet agents (example, aspirin, clopidogrel, coumadin, heparin, or warfarin) that cannot be held to permit tumor biopsy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (22):
- United States (9):
  - UCSD, La Jolla, California
  - Emory, Atlanta, Georgia
  - Massachusetts General, Boston, Massachusetts
  - Barbara Ann Karmanos, Detroit, Michigan
  - Roswell Park, Buffalo, New York
  - Fox Chase, Philadelphia, Pennsylvania
  - Vanderbilt, Nashville, Tennessee
  - Mary Crowley Research Centers, Dallas, Texas
  - US Oncology, Fairfax, Virginia
- Italy (5):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) S.r.l, Meldola
  - Istituto di Ricovero e Cura a Carattere Scientifico - Istituto Clinico Humanitas (Humanitas Research, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero - Universitaria di Modena Policlinico, Modena
  - Azienda Ospedaliera Universitaria Senese - Policlinico Santa Maria Alle Scotte, Siena
- Spain (6):
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Consejo Superior de Investigaciones Cientificas (CSIC) - Centro de Investigacion del Cancer (CIC), Salamanca
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario de Valencia (CHUV), Valencia
- United Kingdom (2):
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital - Northern Centre for Canc, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Juric D, Barve M, Vaishampayan U, Roda D, Calvo A, Janez NM, Trigo J, Greystoke A, Harvey RD, Olszanski AJ, Opyrchal M, Spira A, Thistlethwaite F, Jimenez B, Sappal JH, Kannan K, Riley J, Li C, Li C, Gregory RC, Miao H, Wang S. A phase Ib study evaluating the recommended phase II dose, safety, tolerability, and efficacy of mivavotinib in combination with nivolumab in advanced solid tumors. Cancer Med. 2024 Mar;13(5):10.1002/cam4.6776. doi: 10.1002/cam4.6776. PMID 38501219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in the United States, Spain and United Kingdom from 12 August 2016 to 30 November 2018.
Pre-assignment Details: Participants with advanced solid tumors and metastatic TNBC were enrolled in Parts 1 and 2 respectively. Part 2 cohorts: TNBC cohort was discontinued due to insufficient efficacy of drug. Study was terminated before start of potential fixed dose cohort, non-small cell lung cancer cohort and head and neck squamous cell carcinoma cohort.
Groups:
- Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg: TAK-659 60 milligram (mg), tablets, orally, once daily in each 28-days treatment cycle in combination with nivolumab 3 milligram per kilogram (mg/kg), infusion over 60 minutes, intravenously, on Days 1 and 15 in each 28-days treatment cycle until progressive disease (PD) or unacceptable toxicity (up to Week 48) in Dose Escalation Phase.
- Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg: TAK-659 80 mg, tablets, orally, once daily in each 28-days treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Days 1 and 15 in each 28-days treatment cycle until PD or unacceptable toxicity (up to Week 48) in Dose Escalation Phase.
- Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg: TAK-659 100 mg, tablets, orally, once daily in each 28-days treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Days 1 and 15 in each 28-days treatment cycle until PD or unacceptable toxicity (up to Week 48) in Dose Escalation Phase.
- Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC): TAK-659 80 mg, tablets, orally, once daily in each 28-days treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Days 1 and 15 in each 28-days treatment cycle until PD or unacceptable toxicity (up to Week 13) in Dose Expansion Phase in participants with metastatic triple negative breast cancer (TNBC).
Period: Dose Escalation Phase
Arm/Group | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Started | 8 | 11 | 5 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 8 | 11 | 5 | 0
Not completed — Study Terminated by Sponsor | 1 | 2 | 0 | 0
Not completed — Death | 5 | 6 | 5 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0
Period: Dose Expansion Phase
Arm/Group | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Started | 0 | 0 | 0 | 17
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 17
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 7
Not completed — Death | 0 | 0 | 0 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all the participants who received at least 1 dose of study drug.
Groups:
- Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg: TAK-659 60 mg, tablets, orally, once daily in each 28-days treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Days 1 and 15 in each 28-days treatment cycle until PD or unacceptable toxicity (up to Week 48) in Dose Escalation Phase.
- Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC): TAK-659 80 mg, tablets, orally, once daily in each 28-days treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Days 1 and 15 in each 28-days treatment cycle until PD or unacceptable toxicity (up to Week 13) in Dose Expansion Phase in participants with metastatic TNBC.
- Total: Total of all reporting groups
Arm/Group | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC) | Total
Number analyzed (Participants) | 8 | 11 | 5 | 17 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (8.53) | 51.2 (16.04) | 56.8 (16.22) | 49.2 (8.62) | 52.3 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 2 | 17 | 32
  Male | 3 | 3 | 3 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 10 | 4 | 15 | 37
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2 | 4
  White | 7 | 9 | 4 | 12 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 0 | 0 | 0 | 9 | 9
  United Kingdom | 0 | 0 | 0 | 2 | 2
  United States | 8 | 11 | 5 | 6 | 30
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 166.09 (11.473) | 166.58 (11.360) | 167.00 (5.523) | 164.03 (8.245) | 165.48 (9.334)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 71.75 (19.006) | 60.11 (17.393) | 73.62 (13.646) | 69.50 (12.266) | 67.92 (15.572)

OUTCOME MEASURES:

1. Primary Outcome: Part 1, Dose Escalation Phase: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the dose range at which less than or equal to (<=) 1 of 6 evaluable participants experience dose limiting toxicities (DLT) within the first 28 days of treatment (end of Cycle 1). Toxicities were evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Time Frame: At end of Cycle 1 Day 28
Population: The DLT-evaluable population was defined as participants who had met the minimum treatment and safety evaluation requirements of the study and/or who experienced a DLT during Cycle 1.
Measure: Number; unit: mg
Groups:
- Part 1: Dose Escalation Participants: TAK-659 60 mg, 80 mg or 100 mg, tablets, orally, once daily in each 28-days treatment cycle in combination with nivolumab 3 mg/kg, infusion over 60 minutes, intravenously, on Days 1 and 15 in each 28-days treatment cycle until PD or unacceptable toxicity (up to Week 48).
Arm/Group | Part 1: Dose Escalation Participants
Number analyzed (Participants) | 19
mg | 80

2. Primary Outcome: Part 1, Dose Escalation Phase: Recommendation Phase 2 Dose (RP2D)
Description: RP2D was evaluated from cumulative toxicities in Cycle 1 and beyond. Toxicities were evaluated according to NCI CTCAE version 4.03.
Time Frame: Up to Cycle 12 (each Cycle length is equal to [=] 28 days)
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | Part 1: Dose Escalation Participants
Number analyzed (Participants) | 19
mg | 80

3. Primary Outcome: Part 2, Dose Expansion Phase: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who's best overall response (BOR) was either complete response (CR) or partial response (PR). The ORR assessment was based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The BOR was defined as the best response recorded from the start of the study treatment until the start of subsequent anticancer therapy. CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to less than (<) 10 millimeter (mm). PR: was at least a 30 percent (%) decrease in sum of diameter (SOD) of target lesions, taking as reference the baseline SOD.
Time Frame: From the start of study treatment until the start of subsequent anticancer therapy (up to 28 months)
Population: The response-evaluable population was defined as participants who received at least 1 dose of study drug, had measurable disease at Baseline, and had at least 1 post-baseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Number analyzed (Participants) | 15
percentage of participants | 0

4. Secondary Outcome: Percentage of Participants Who Experienced at Least One Treatment-emergent Adverse Events (TEAEs), Grade 3 or 4 Adverse Events (AEs), Serious Adverse Events (SAEs), and TEAEs Leading to Discontinuation
Description: AEs Grades were evaluated as per NCI CTCAE version 4.03.
Time Frame: From the first dose of the study drug up to 28 days after the last dose of the study drug or the start of subsequent anticancer therapy (up to 28 months)
Population: The safety population was defined as all the participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Number analyzed (Participants) | 8 | 11 | 5 | 17
percentage of participants
  TEAEs | 100 | 100 | 100 | 100
  Grade 3 or 4 AEs | 87.5 | 81.8 | 100 | 76.5
  SAEs | 75.0 | 63.6 | 80.0 | 70.6
  TEAEs Leading to Discontinuation | 25.0 | 27.3 | 20.0 | 23.5

5. Secondary Outcome: Part 2, Dose Expansion Phase: Disease Control Rate (DCR)
Description: DCR was the percentage of participants who had BOR with either CR, PR, or stable disease (SD). The DCR assessment was based on RECIST version 1.1. The BOR was defined as the best response recorded from the start of the study treatment until the start of subsequent anticancer therapy. CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR: was at least a 30% decrease in SOD of target lesions, taking as reference the baseline SOD. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SOD.
Time Frame: From the start of study treatment until the start of subsequent anticancer therapy (up to 28 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Number analyzed (Participants) | 15
percentage of participants | 26.7

6. Secondary Outcome: Part 2, Dose Expansion Phase: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a response to the date of first documented progressive disease. DOR assessment was based on RECIST v1.1. CR: was disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR: at least 30% decrease in SOD of target lesions, taking as reference the baseline SOD. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. DOR was calculated using Kaplan-Meier analysis.
Time Frame: From the date of first documentation of a response to the date of first documented PD (up to 28 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Number analyzed (Participants) | 15
months | NA [NA to NA] — Median, lower and upper limit of confidence interval could not be calculated because no participant had an event.

7. Secondary Outcome: Part 2, Dose Expansion Phase: Percentage of Participants With PD at Month 6
Description: PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. The PD assessment was based on RECIST v1.1.
Time Frame: Month 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Number analyzed (Participants) | 15
percentage of participants | 86.7

8. Secondary Outcome: Part 2, Dose Expansion Phase: Progression Free Survival (PFS)
Description: PFS was defined as the time from date of first study drug administration to the date of first documented PD or death due to any cause, whichever occurred first. The PFS assessment was based on RECIST v1.1. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions. PFS was calculated using Kaplan-Meier estimate.
Time Frame: From the date of first study drug administration up to date of first documented PD or death due to any cause, whichever occurred first (up to 28 months)
Population: The safety population was defined as all the participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Number analyzed (Participants) | 17
months | 1.7 [1.0 to 2.8]

9. Secondary Outcome: Part 2, Dose Expansion Phase: Overall Survival (OS)
Description: OS was calculated from date of participant enrollment to the date of participant's death due to any cause. OS was assessed based on RECIST v 1.1. Participants without documentation of death at time of the analysis were censored as of the date the participant was last known to be alive, or the data cutoff date, whichever was earlier. OS was calculated using Kaplan-Meier estimate. Enrollment was defined as the time of the initiation of the first dose of study drug.
Time Frame: Baseline up to the date of death due to any cause (up to 28 months)
Population: The safety population was defined as all the participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
Number analyzed (Participants) | 17
months | 4.9 [3.1 to NA] — Upper Limit of confidence interval could not be estimated due to insufficient number of events.

10. Secondary Outcome: Part 1, Dose Escalation Phase, Cmax: Maximum Observed Plasma Concentration for TAK-659
Time Frame: Cycle 1, Days 1 and 15: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: The pharmacokinetic (PK)-evaluable population was defined as participants with sufficient concentration-time and dosing data to reliably estimate PK parameters. PK-evaluable population where data at specified time points was available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 8 | 11 | 5
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 84.02 (56.11) | 212.51 (64.69) | 165.60 (55.53)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 8 | 3
  Cycle 1 Day 15 | 132.04 (67.98) | 236.08 (58.99) | 379.82 (26.66)

11. Secondary Outcome: Part 1, Dose Escalation Phase, Tmax: Time to Reach the Cmax for TAK-659
Time Frame: Cycle 1, Days 1 and 15: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: The PK-Evaluable population was defined as participants with sufficient concentration-time and dosing data to reliably estimate PK parameters. PK-evaluable population where data at specified time points was available.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 8 | 11 | 5
hour
  Cycle 1 Day 1 | 2.2000 [0.417 to 7.500] | 2.0667 [0.500 to 4.100] | 3.7000 [0.900 to 4.050]
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 8 | 3
  Cycle 1 Day 15 | 1.9833 [1.117 to 4.033] | 3.8583 [2.000 to 5.017] | 3.8333 [2.050 to 3.967]

12. Secondary Outcome: Part 1, Dose Escalation Phase, AUCtau: Area Under the Plasma Concentration-time Curve From Time 0 to Tau Over the Dosing Interval for Area Under the Plasma Concentration for TAK-659
Time Frame: Cycle 1, Days 1 and 15: pre-dose and at multiple time points (up to 24 hours) post-dose (Cycle length= 28 days)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg
Number analyzed (Participants) | 8 | 11 | 5
hour*nanogram per milliliter (h*ng/mL)
  Cycle 1 Day 1 | 845.7076 (24.5906) | 1867.3673 (59.4921) | 1745.0750 (56.3522)
  Cycle 1 Day 15: number analyzed (Participants) | 4 | 6 | 3
  Cycle 1 Day 15 | 1906.1855 (28.4065) | 2259.5453 (35.4104) | 4515.3938 (37.5764)

ADVERSE EVENTS:
Time Frame: TEAEs are AEs that started after the first dose of study drug and no more than 28 days after the last dose of study drug (up to 28 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Reported AEs and deaths are TEAEs that occurred between the first dose of the study drug and 28 days after the last dose of the study drug.
Arm/Group | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC)
All-Cause Mortality (participants affected / at risk) | 5/8 | 6/11 | 5/5 | 8/17
Serious Adverse Events (participants affected / at risk) | 6/8 | 7/11 | 4/5 | 12/17
Other Adverse Events (participants affected / at risk) | 8/8 | 11/11 | 5/5 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg (N=8) | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg (N=11) | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg (N=5) | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC) (N=17)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (5)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: TAK-659 60 mg + Nivolumab 3 mg/kg (N=8) | Part 1: TAK-659 80 mg + Nivolumab 3 mg/kg (N=11) | Part 1: TAK-659 100 mg + Nivolumab 3 mg/kg (N=5) | Part 2: TAK-659 80 mg + Nivolumab 3 mg/kg (TNBC) (N=17)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 7 (21) | 1 (1) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (5) | 8 (13) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 4 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (1) | 3 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 2 (4) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (9) | 4 (4) | 3 (4) | 5 (7)
Pyrexia (General disorders) | 2 (4) | 3 (4) | 2 (6) | 6 (8)
Oedema peripheral (General disorders) | 3 (4) | 2 (5) | 0 (0) | 5 (6)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 6 (16) | 4 (5) | 7 (10)
Alanine aminotransferase increased (Investigations) | 2 (3) | 6 (10) | 3 (3) | 5 (6)
Amylase increased (Investigations) | 0 (0) | 6 (12) | 3 (4) | 4 (6)
Lipase increased (Investigations) | 0 (0) | 5 (9) | 3 (7) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (13)
Troponin increased (Investigations) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (3) | 2 (2) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram ST-T segment abnormal (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood corticotrophin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transferrin saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 6 (9) | 2 (2) | 6 (6)
Nausea (Gastrointestinal disorders) | 5 (7) | 2 (2) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (5) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (9) | 4 (6) | 1 (1) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 1 (1) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 6 (7) | 1 (1) | 3 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 4 (7)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Resting tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (5) | 6 (9) | 2 (7) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (3) | 0 (0) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (3) | 2 (3) | 4 (12)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exophthalmos (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Testicular oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT02834247/Prot_001.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT02834247/SAP_000.pdf